CLINICAL TRIAL: NCT04467021
Title: Cancer Therapy Risk-Reduction With Intensive Systolic BP Management (CARISMA) - a Phase II Study
Brief Title: Cancer and Blood Pressure Management, CARISMA Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ECOG-ACRIN Cancer Research Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: Eastern Cooperative Oncology Group (Network)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EAQ191; NCI-2020-00900 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); EAQ191 (Other: ECOG-ACRIN Cancer Research Group); ECOG-ACRIN-EAQ191 (Other: DCP); EAQ191 (Other: CTEP); UG1CA189828 (NIH)
Record Dates: First submitted 2020-07-07; First posted 2020-07-10 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Cardiovascular Disorder; Chronic Kidney Disease; Metastatic Renal Cell Carcinoma; Metastatic Thyroid Gland Medullary Carcinoma; Stage IV Renal Cell Cancer AJCC v8; Stage IV Thyroid Gland Medullary Carcinoma AJCC v8; Stage IVA Thyroid Gland Medullary Carcinoma AJCC v8; Stage IVB Thyroid Gland Medullary Carcinoma AJCC v8; Stage IVC Thyroid Gland Medullary Carcinoma AJCC v8
MeSH Terms: conditions — Cardiovascular Diseases; Renal Insufficiency, Chronic; Carcinoma, Renal Cell; Carcinoma, Medullary | interventions — Practice Guidelines as Topic; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (intensive systolic blood pressure management) (Experimental): Patients receive intensive systolic blood pressure management for 6 months. Patients receive increased blood pressure medication every 2 weeks while systolic blood pressure is 120 mmHg or higher. Patients also monitor blood pressure at home 1 day a week (4 times in 1 day) every 2 weeks, and upload the recorded blood pressure readings to the provider and to a central blood pressure monitoring team. Patients with changes in blood pressure medications monitor blood pressure readings on 3 days in 1 week (4 times in 1 day).
  Interventions: Other: Blood Pressure Measurement; Other: Clinical Management; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Arm B (usual blood pressure management) (Active Comparator): Patients receive standard blood pressure management for 6 months. Patients receive blood pressure medications per doctor's instruction. Patients also monitor blood pressure at home 1 day (4 times in 1 day) every 2 weeks, and upload the recorded blood pressures to a central monitoring team.
  Interventions: Other: Best Practice; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Other: Best Practice — Receive usual blood pressure management
  Other Names: standard of care; standard therapy
  Arms: Arm B (usual blood pressure management)
Other: Blood Pressure Measurement — Undergo blood pressure measurement
  Arms: Arm A (intensive systolic blood pressure management)
Other: Clinical Management — Undergo intensive systolic BP management
  Arms: Arm A (intensive systolic blood pressure management)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase II trial studies how well intensive blood pressure management works in decreasing systolic blood pressure in patients with kidney or thyroid cancer that has spread to other places in the body (metastatic) who are starting anti-angiogenic tyrosine kinase inhibitor cancer therapy. This study is being done to find out if a systolic blood pressure to a target of less than 120 mmHg (intensive systolic blood pressure management) can be achieved, well tolerated, and beneficial as compared to the usual approach to a target of less than 140 mmHg while taking an anti-angiogenic tyrosine kinase inhibitor. This study may help doctors understand the best way to control blood pressure in kidney or thyroid cancer patients taking anti-angiogenic tyrosine kinase inhibitor.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the feasibility of an intensive (systolic blood pressure [SBP] < 120 mmHg) "Intervention" versus standard care (SBP < 140 mmHg) "Non-Intervention" approach to blood pressure (BP) control in metastatic renal cell and thyroid cancer patients initiating anti-angiogenic tyrosine kinase inhibitors.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM A: Patients receive intensive systolic blood pressure management for 6 months. Patients receive increased blood pressure medication every 2 weeks while systolic blood pressure is 120 mmHg or higher. Patients also monitor blood pressure at home 1 day a week (4 times in 1 day) every 2 weeks and upload the recorded blood pressure readings to the provider and to a central blood pressure monitoring team. Patients with changes in blood pressure medications monitor blood pressure readings on 3 days in 1 week (4 times in 1 day).

ARM B: Patients receive standard blood pressure management for 6 months. Patients receive blood pressure medications per doctor's instruction. Patients also monitor blood pressure at home 1 day (4 times in 1 day) every 2 weeks and upload the recorded blood pressures to a central monitoring team.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* Patient must have histologically or cytologically-proven advanced metastatic renal cell cancer (mRCC) or medullary thyroid cancer initially treated with anti-angiogenic tyrosine kinase inhibitors (AA-TKIs) including: sunitinib, sorafenib, pazopanib, cabozantinib, lenvatinib, vandetanib, or axitinib)

  * NOTE: If patient has a severe sulfa allergy (e.g. Stevens Johnson reaction), then alternative non-sulfa medications can be considered in consultation with the C-BAC. Patient with a noted severe allergic reactions to medications listed in the algorithms is not necessarily excluded from this trial, as alternative medications could be considered in consultation with the C-BAC. Moreover, the patient treated with pre-existing medications that may interact with proposed BP medications is not necessarily excluded, as alternative medications exist. The clinical significance of any potential drug interactions can also be addressed with the C-BAC.
* Prior exposure to another AA-TKI is permissible. Concurrent or prior treatment with immunotherapy is also permissible
* Patient must have either clinical cardiovascular (CV) disease or evidence of increased CV risk as defined by one or more of the following:

  * Clinical CV disease (history of myocardial infarction [MI] acute coronary syndrome, coronary revascularization, carotid endarterectomy or stenting greater than 3 months prior to registration, peripheral artery disease, cerebrovascular accident greater than 3 months prior to registration, abdominal aortic aneurysm or heart failure [HF])
  * An American College of Cardiology/American Heart Association (ACC/AHA) CV risk score of at least 10%
  * Chronic kidney disease (defined as an estimated glomerular filtration rate [eGFR] between 30 and 60 ml/min per 1.73 m^2). Dialysis patients and patients with an eGFR < 30 ml/min/1.73m^2 will be excluded. eGFR will be calculated according to the Chronic Kidney Disease Epidemiology Collaboration (CKD-Epi) equation
* Patient must have systolic blood pressure (SBP) >= 130 mmHg on two or more occasions according to any in-clinic visit in the 12 weeks prior to or during their initial 4 weeks of treatment with an AA-TKI. Patient who have a prior diagnosis of hypertension or on pre-existing anti-hypertensive medications are eligible for enrollment. However, patient must not be on more than 3 baseline blood pressure medications at time of entry

  * NOTE: If a patient has a single elevated SBP >= 130mmHg but not on repeat assessment, an additional SBP assessment should be performed to confirm ineligibility
* Patient must agree to comply with performing home blood pressure monitoring using an Omron7250 oscillometric monitor at home, or equivalent models
* Women of childbearing potential and sexually active males must be strongly advised to use accepted and effective methods of contraception or to abstain from sexual intercourse for the duration of their participation in the study
* Patient must have internet access through a computer, tablet, or smart phone to use EASEE-PRO and home BP monitoring. A valid phone number to receive text messages and email address are also necessary
* Leukocytes >= 3,000/mcL (obtained within 14 days prior to registration)
* Absolute neutrophil count >= 1,500/mcL (obtained within 14 days prior to registration)
* Platelets >= 100,000/mcL (obtained within 14 days prior to registration)
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional upper limit of normal (ULN) (obtained within 14 days prior to registration)
* Patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
* Patient with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* Patient with treated brain metastases are eligible if follow-up brain imaging after central nervous system (CNS)-directed therapy shows no evidence of progression
* Patient with new or progressive brain metastases (active brain metastases) or leptomeningeal disease are eligible if the treating physician determines that immediate CNS specific treatment is not required and is unlikely to be required during the first cycle of therapy
* Patient with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* Patient must have an Eastern Cooperative Oncology Group (ECOG) performance status 0-2

Exclusion Criteria:

* Patient must not have end-stage renal failure on dialysis, history of repeated hyperkalemia with a potassium > 5.5 mEq/l, or have a kidney transplant, or an eGFR < 30 ml/min/1.73 m^2
* Patient must not have coronary artery bypass grafting, MI acute coronary syndrome severe/unstable angina, stroke, transient ischemic attack, clinically significant bleeding requiring hospitalization or pulmonary embolism within 3 months prior to registration
* Patient must not have brain surgery or radiotherapy within 2 weeks prior to registration
* Patient must not have uncontrolled blood pressure defined by SBP > 160 mmHg on three or more antihypertensives prior to TKI initiation
* Patient with an arm circumference too large (> 50 cm) or small (< 17 cm) to allow accurate BP measurement with available devices will not be eligible
* Women must not be pregnant or breast-feeding due to the potential harm to an unborn fetus and possible risk for adverse events in nursing infants with some anti-hypertensives, including angiotensin receptor blockers. All females of childbearing potential must have a blood test or urine study within 14 days prior to registration to rule out pregnancy. A female of childbearing potential is defined as any woman, regardless of sexual orientation or whether they have undergone tubal ligation, who meets the following criteria: has achieved menarche at some point, has not undergone a hysterectomy or bilateral oophorectomy; or has not been naturally postmenopausal (amenorrhea following cancer therapy does not rule out childbearing potential) for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2020-10-29 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Differences in systolic blood pressure (SBP) based on automated office BP measurements | Up to 6 months
  Differences in SBP over the 6- month study period between intensive BP control (intervention) versus standard care (non-intervention group) will be compared using the "difference-indifference" method. All mixed effects models will be estimated using generalized estimating equations (GEE).

SECONDARY OUTCOMES:
Difference in SBP based on all automated home and office BP measurements | Up to 6 months
  Based on all automated home and office BP measurements.
Study retention rates | Up to 6 months
  Will compare the study retention rates between the intensive SBP versus standard care group, by constructing appropriate mixed-effect generalized linear models (e.g. a mixed effect log-linear model for fatigue and a logistic model for study retention) and using GEE for model estimation
Frequency of automated home SBP measurements > 180 mmHg or < 90 mmHg or diastolic (D)BP > 110 mmHg | Up to 6 months
  The frequency of orthostatic hypotension as defined by > 20 mmHg decreases in office SBP with standing; or symptomatic hypotension, as defined by the Common Terminology Criteria for Adverse Events (CTCAE) criteria, in participants in the intervention and non-intervention group arms.
Differences in symptoms and health-related quality of life | Up to 6 months
  Will compare the Patient Reported Outcomes Measurement Information System (PROMIS) Fatigue between the intensive SBP versus standardlcCare group, by constructing appropriate mixed-effect generalized linear models (e.g. a mixed effect log-linear model for fatigue and a logistic model for study retention) and using GEE for model estimation.
Differences in patient-reported medication compliance | Up to 6 months
  Will compare the medication compliance between the intensive SBP versus standard care group, by constructing appropriate mixed-effect generalized linear models (e.g. a mixed effect log-linear model for fatigue and a logistic model for study retention) and using GEE for model estimation.
Patient-rated adverse events associated with hypertension, hypotension and anti-hypertensive medications | Up to 6 months
Participant satisfaction with BP care | Up to 6 months
  The participant satisfaction with BP care (including the C-BAC and the related technologies) and BP medications will be evaluated through questionnaires evaluated on a Likert scale and via open ended discussions with focus groups.
Provider satisfaction with BP care | Up to 6 months
  The provider satisfaction with BP care (including the C-BAC and the related technologies) and BP medications will be evaluated through questionnaires evaluated on a Likert scale and via open ended discussions with focus groups.

OTHER OUTCOMES:
Incidence of significant cardiovascular (CV) events | Up to 6 months
  Will determine the rates of adverse cardiovascular events in each group. These include the incidence of significant CV events including stroke, acute coronary syndrome/myocardial infarction or hospitalization for heart failure; the suspension of anti-angiogenic tyrosine kinase inhibitors therapy due to toxicity; or all-cause death.

CONTACTS AND LOCATIONS:
Overall Officials: Bonnie Ky, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (25):
- United States (25):
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center-Weiler Hospital, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Aurora Saint Luke's South Shore, Cudahy, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin

REFERENCES:
- [Derived] Narayan V, Liu T, Song Y, Mitchell J, Sicks J, Gareen I, Sun L, Denduluri S, Fisher C, Manikowski J, Wojtowicz M, Vadakara J, Haas N, Margulies KB, Ky B. Early Increases in Blood Pressure and Major Adverse Cardiovascular Events in Patients With Renal Cell Carcinoma and Thyroid Cancer Treated With VEGFR TKIs. J Natl Compr Canc Netw. 2023 Oct;21(10):1039-1049.e10. doi: 10.6004/jnccn.2023.7047. PMID 37856199